CLINICAL TRIAL: NCT03467984
Title: A Single-blind, Multi-center, Randomized, Active-controlled, Parallel Group, Phase II Study to Evaluate the Safety and Immunogenicity of Intramuscular Three Injections With LBVE(Multivalent Pneumococcal Conjugate Vaccine) Compared to Prevnar13 in Healthy Infants
Brief Title: A Study to Evaluate the Safety and Immunogenecity of LBVE(Multivalent Pneumococcal Conjugate Vaccine) in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LG-VECL002
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBVE (Experimental): Infants will receive a 0.5mL intramuscular injection of LBVE at 6,10 and 14 weeks of age
  Interventions: Biological: LBVE
- Prevnar13 (Active Comparator): Infants will receive a 0.5mL intramuscular injection of Prevnar13 at 6,10 and 14 weeks of age
  Interventions: Biological: Prevnar13

INTERVENTIONS:
Biological: LBVE — Multivalent pneumococcal conjugate vaccine be administered by Intramuscular injection into the thigh
  Arms: LBVE
Biological: Prevnar13 — 13-valent pneumococcal conjugate vaccine be administered by Intramuscular injection into the thigh
  Arms: Prevnar13

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of LBVE (Multivalent Pneumococcal Conjugate Vaccine) in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants of either sex who have reached at least 42 days (6 weeks) of age and not more than 56 days (8 weeks) of age at the time of enrollment.
* The parents or LAR(Legally authorized representative) able to understand and comply with planned study procedures.
* Signed informed consent by subject's parents or LAR(Legally authorized representative)

Exclusion Criteria:

* Previously received any pneumococcal vaccine
* Receipt of immunoglobulin or blood-derived product before the study
* Known or suspected immune disorder, or received immunosuppressive therapy
* Known major congenital malformation or serious chronic disorder
* Participation in another interventional trial

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving pneumococcal serotype-specific IgG >= 0.35 ug/ml | 4 weeks after 3rd(last) vaccination
Pneumococcal serotype-specific IgG geometic mean concentration (GMC) ratios | 4 weeks after 3rd(last) vaccination

SECONDARY OUTCOMES:
Proportion of subjects achieving targeted pneumococcal serotype-specific opsonophagocytic assay (OPA) titer | 4 weeks after 3rd(last) vaccination
Pneumococcal serotype-specific OPA geometic mean titer (GMT) ratios | 4 weeks after 3rd(last) vaccination
Solicited adverse events | Baseline(pre-vaccination) up to 7 days after each vaccination
Unsolicited adverse events | Baseline(pre-vaccination) up to 4 weeks after 3rd(last) vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- LG chem, Seoul, Gangseo-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No